CLINICAL TRIAL: NCT00824694
Title: Impact of Accu-Chek 360 View on Practice Patterns and HBA1C in Veterans With Type 2 Diabetes.
Brief Title: Impact of Accu-Chek 360 in Veterans With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomedical Research Institute of New Mexico (Other)
Collaborators: New Mexico VA Healthcare System (U.S. Federal Agency); Carl T. Hayden VA Medical Center (U.S. Federal Agency); Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Glen H. Murata, M.D., New Mexico VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Investigator Initiated
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes
Keywords: Glucose; Diabetes Mellitus, Type 2; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): The intervention will consist of targeted SMBG, provider training and patient education-all of which are focused on normalizing the most significant glucose abnormalities at any given time. SMBG will alternate between 2 strategies: glucose profiling and target monitoring. Intervention PCP's will use 380 View to identify a patient's most significant glucose elevations(s) and devise a treatment plan that includes drug type, dose increases, monitoring times, goal for the target, and stop criteria.
  Interventions: Other: Targeted Self-Monitoring Of Blood Glucose (SMBG); Other: Provider Training; Other: Patient Education
- Control Arms (Active Comparator): Subjects will repeat the dose titration cycle under the guidance of a case manager until the target is reached, maximal recommended doses of medications are used, or a stop criterion is met. They will then resume glucose profiling to identify the next target. This process is repeated until all targets reach their optimal value. Control patients will monitor and be treated in the customary manner.
  Interventions: Other: Targeted Self-Monitoring Of Blood Glucose (SMBG); Other: Provider Training; Other: Patient Education

INTERVENTIONS:
Other: Targeted Self-Monitoring Of Blood Glucose (SMBG) — SMBG will alternate between 2 strategies: glucose profiling and target monitoring.
Other: Provider Training — Focused on normalizing the most significant glucose abnormalities at any given time.
Other: Patient Education — Focused on normalizing the most significant glucose abnormalities at any given time.

SUMMARY:
To show that a structured treatment plan based upon Accu-Chek 360 View has a favorable effect on physician decision-making and HbA1c for patients on oral hypoglycemic agents (OHA) or insulin for type 2 diabetes (T2D).

Hypothesis 1: Compared to controls, intervention subjects will undergo a greater number of medication changes and have a lower HbA1 at the conclusion of the study.

Hypothesis 2: Higher rates of monitoring at entry will be associated with lower CHO consumption, lower percent body fat, higher medication compliance, and higher physical activity levels.

Hypothesis 3: Patients with lower rates of monitoring at entry will have higher rates of depression, more likely to have an external locus of control, and express greater fear about self-testing.

DETAILED DESCRIPTION:
Primary care providers (PCP's) will be randomized to intervention and control arms. Their T2D patients will be identified by searching computerized pharmacy records for OHA or insulin, followed until they are on a stable medical regimen, and eligible to participate if their baseline HbA1c is 7.0 - 9.5% if on OHA or 7.5 - 10.0% if on insulin. Two sample frames will be created for intervention patients: one of patients on OHA alone and one of patients on insulin alone or in combination with OHA. The same procedure will be used to develop corresponding sample frames for control patients. OHA patients will be randomly sampled from the intervention and control groups at a ratio of 1:1 until 174 subjects have been enrolled. Insulin patients will be recruited in the same manner until another 174 subjects are recruited. At entry, patients will have measurements of fat mass, insulin-resistance, stimulated C-peptide, carbohydrate intake, and physical activity level.

The intervention will consist of targeted SMBG, provider training, and patient education, all of which will be focused on normalizing the most significant glucose abnormalities at any given time. SMBG will alternate between 2 strategies: glucose profiling and target monitoring. Intervention PCP's will use 360 View to identify a patient's most significant glucose elevation(s) and devise a treatment plan that includes the medication to be used, starting dose, dose increment per cycle, interval between dose increases, monitoring times and frequency, goal for the target, and stop criteria. Separate treatment protocols will be recommended for OHA patients with basal hyperglycemia, OHA patients with PP hyperglycemia, insulin patients with basal hyperglycemia, and insulin patients with PP hyperglycemia. Treatment will conform to current standards of practice as defined by package inserts and Micromedex, the VA's official on-line drug reference. Subjects will repeat the dose titration cycle under the guidance of a case manager until the target is reached, maximal recommended doses of medications are used, or a stop criterion is met. They will then resume glucose profiling to identify the next target. This process is repeated until all targets reach their optimal value. Intervention subjects will undergo no less than 4 cycles in 48 weeks. Control patients will monitor and be treated in the customary manner.

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary care provider
* Diabetes diagnosed after age 35
* Eat 3 meals daily and ≤ 1 snack
* If on OHA, have willingness to start insulin

Exclusion Criteria:

* Type 1 diabetes or DKA
* On insulin pump or CGM
* Preference for language other than English
* Can't or won't monitor
* Unfavorable occupation or living arrangements
* Terminal illness
* Active alcoholism or substance abuse
* Severe depression
* Chronic liver disease
* Pituitary or adrenal dysfunction
* Immunosuppression
* Hct < 35
* Creatinine ≥ 2.5

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Principal endpoints will be measured 48 weeks after group assignment and include the number of medication changes and HbA1c. Interim analysis will include HbA1c measurement at 3 mont intervals. | 48 weeks

SECONDARY OUTCOMES:
Secondary endpoints include changes in patient attitudes toward SMBG, daily carbohydrate consumption, physical activity level, BMI, and medication compliance (for subjects on OHA). | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Glen H Murata, M.D., Principal Investigator — New Mexico VA Healthcare System
Locations (3):
- United States (3):
  - Carl T. Hayden VAMC, Phoenix, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - New Mexico VA Health Care System, Albuquerque, New Mexico